CLINICAL TRIAL: NCT00866164
Title: Prometra's Utilization in Mitigating Pain II
Acronym: (PUMP 2)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Flowonix Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: G060192/S019
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Intractable Pain; Back Pain; Leg Pain; Arm Pain; Trunk Pain
Keywords: back pain; intractable pain; implantable infusion pump; morphine
MeSH Terms: conditions — Pain, Intractable; Back Pain

INTERVENTIONS:
Device: Prometra Programmable Pump — Implantation of Prometra Pump for delivery of intrathecal morphine for the treatment of chronic intractable pain

SUMMARY:
Intrathecal infusion pumps are increasingly used to deliver analgesics for chronic intractable pain. The PUMP II trial is designed to evaluate the ongoing safety and efficacy of the new Prometra® Programmable Pump System for intrathecal administration of morphine sulfate to treat chronic intractable pain.

DETAILED DESCRIPTION:
The development of fully implantable systems changed the dynamics and risks associated with intrathecal drug delivery. Pump reservoirs could be refilled with medication more infrequently (every 1-3 months), greatly reducing the risk of infection. Pumps were initially driven by the pressure differential of an injected gas, pushing drug at a fixed rate from an isolated chamber through an orifice of predetermined size. Later, mechanical pumps were developed that allowed for programmability of different infusion rates, and complex administration of infusions and preset boluses. These pumps have dominated the US market for long-term intrathecal drug delivery systems (IDDSs), and have expanded the range of conditions and patients that can be treated successfully.

Because IDDSs characteristically deliver low flow rates of drug to the intrathecal space (<1 mL/day), the reliability, durability, and accuracy of the pump are critical for the efficacy and safety of treatment. This continued access trial will assess the ongoing safety and efficacy of a new fully implanted IDDS, the Prometra Programmable Pump.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is suffering from cancer pain requiring strong opioids (e.g., fentanyl, methadone, levorphanol, hydromorphone, oxymorphone, oxycodone) OR Patient has chronic, non-malignant pain OR Patient needs an implantable pump system (pump AND catheter) replaced due to malfunction or battery depletion. Patient must have documented history of sufficient pain relief with intrathecal morphine sulfate infusion.
2. Patient is 18 years of age or older.
3. Patient has life expectancy of > 6 months.
4. Patient has documented failure to respond to less invasive methods of pain control, including attempts to eliminate physical and behavioral abnormalities that may cause an exaggerated reaction to pain.
5. Patient has pain that is ineffectively controlled by single or multiple systemic (oral, rectal, transdermal or intravenous) analgesic treatments or patient experienced intolerable side effects from such treatment.
6. Patient has had a successful trial of morphine sulfate (intrathecal or epidural) for relief of the target symptoms.
7. Patient agrees to obtain pain medication prescriptions only from the investigator.
8. Patient has provided written informed consent to participate in the study.
9. Patient is considered by the investigator to be a medically and psychologically appropriate candidate for pump implantation.
10. Investigator and/or study coordinator considers the patient to be able and willing to fulfill all study requirements.

Exclusion Criteria:

1. Patient has existing damage to the spinal column observed via MRI of spine that, in the opinion of the Investigator, would prevent intraspinal drug administration (e.g. cord compression from metastatic tumor that could obstruct catheter placement or drug flow). If the patient has a medical condition that contraindicates MRI, the investigator should proceed with the closest appropriate study (i.e. CT scan, X-ray) to rule out any spinal abnormalities that would prevent intraspinal drug administration.
2. Patient has a systemic infection that, in the opinion of the investigator, contraindicates an implantable pump.
3. Patient's anatomy is not large enough to accommodate the pump's size and weight.
4. Patient is pregnant or breast-feeding or is of child-bearing potential and not employing effective birth control.
5. Patient has known allergies or sensitivities to pump system materials (e.g., silicone rubber, titanium, polyphenylsulfone, acetal resin, polyvinylidene fluoride, tungsten).
6. Patient has known allergies to morphine or would be contraindicated for morphine, based on the drug labeling.
7. Patient has a major coexisting medical condition (such as gastrointestinal problems, respiratory reserve / lung function problems, or heart conditions that cannot tolerate further lowering of blood pressure) that, in the opinion of the investigator, contraindicates an implantable pump.
8. Patient will require MRI evaluation post-implantation.
9. Patient has other implanted cardiac electronic devices.
10. Patient has an occupation where he/she would be exposed to high current industrial equipment, powerful magnets or transmitting towers, such as, electricians, electrical engineers or MRI technicians.
11. Patient is unable to participate in all necessary study activities due to physical or mental limitations.
12. Patient is unable or unwilling to return for all required follow-up visits.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult